CLINICAL TRIAL: NCT00004135
Title: Allogeneic Stem Cell Transplantation of Renal Cell Cancer and Metastatic Melanoma After Non-Myeloablative Chemotherapy
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Melanoma or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9672; UCCRC-9672; UCCRC-CTRC-9866; NCI-G99-1612
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — Filgrastim; Cyclophosphamide; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Fludarabine 30 mg/m2/d x S days IVPB in 100 cc NS over 30 minutes on day -8, -7, -6, -S, and -4. Cyclophosphamide 2 gm/m2/d x 2 days IVPB in SOO cc DS W over I hour on day -3 and day-2. G-CSF (Neupogen®) administration 480 f!gld subcutaneously starting on day +5 (or first day of neutropenia if earlier)and continued until an ANC of 0.5 x 109/L is maintained for 3 consecutive days.
  Interventions: Biological: filgrastim; Biological: therapeutic allogeneic lymphocytes; Drug: cyclophosphamide; Drug: fludarabine phosphate; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus peripheral stem cell transplantation in treating patients who have metastatic kidney cancer or melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the safety of nonmyeloablative chemotherapy followed by allogeneic peripheral blood stem cell transplantation in patients with metastatic renal cell carcinoma or melanoma.
* Determine the incidence and severity of all adverse events related to this treatment regimen in this patient population.
* Determine the efficacy of this treatment regimen in terms of tumor regression, response duration, progression free survival, and overall survival in these patients.
* Measure the resulting chimerism and immune reconstitution in these patients after this treatment regimen and correlate with clinical response.

OUTLINE: Patients receive fludarabine IV over 30 minutes on days -8 through -4 and cyclophosphamide IV over 1 hour on days -3 and -2. Immediately following each daily donor leukapheresis, patients receive allogeneic peripheral blood stem cells (PBSC) IV over 15 minutes beginning on day 0 and continuing until the target cells are collected. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 5 and continuing until blood counts recover.

If no graft versus host disease has developed within 4 weeks of allogeneic PBSC transplantation, patients with disease progression or recurrence who have residual donor hematopoiesis on chimerism analysis may receive donor T lymphocytes IV over 30 minutes. Patients may receive an additional course of donor T lymphocytes at the investigator's discretion.

Patients are followed at days 30 and 100, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 10-38 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma or melanoma that is not potentially curable by surgery
* Evaluable disease or bidimensionally measurable disease on physical examination, chest x-ray, CT scan, or MRI

  * Measurable disease by radiography must be reproducible
  * Bony disease or effusions not measurable
* No active CNS disease currently receiving radiotherapy or steroids
* No effusion or ascites of more than 1 liter prior to drainage
* HLA 5/6 or 6/6 matched sibling donor available

  * No known hypersensitivity to E. coli derived products
  * No active infection
  * No health condition that would preclude donation

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* CALGB 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 g/dL
* No active hepatitis

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* LVEF at least 50%

Pulmonary:

* DLCO at least 50% of predicted

Other:

* No active infection
* HIV negative
* No psychological problem that would preclude study compliance
* No known hypersensitivity to E. coli derived products
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior systemic chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1999-02; Primary Completion 2004-10 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Zimmerman, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States